CLINICAL TRIAL: NCT03337607
Title: A Prospective, Randomized, Controlled, Single Centre Trial to Assess the Efficacy and Safety of Radial Extracorporeal Shock Wave Therapy in Patients With Chronic Non-specific Low Back Pain
Brief Title: Radial Extracorporeal Shock Wave Therapy for Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FengDolorClastLowBackPain
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
Keywords: Extracorporeal shock wave therapy; ESWT; Radial extracorporeal shock wave therapy; rESWT; Chronic non-specific low back pain; Non-steroidal anti-inflammatory drug
MeSH Terms: conditions — Low Back Pain | interventions — Celecoxib; Anti-Inflammatory Agents, Non-Steroidal; eperisone; Parasympatholytics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A medical assistant at the Department of Pain Medicine at the First Affiliated Hospital of Zhejiang University will allocate interventions by means of opaque sealed envelopes that will be marked according to the allocation schedule. The medical assistant will be unaware of the size of the blocks.
  The randomized intervention assignment as outlined above will be concealed from both patients and health care staff until recruitment will be complete and irrevocable.
  Neither patients nor therapists will be blinded in the proposed study. The therapist will be the person who will administer rEWST to the patient.
  The assessor will be blinded in the proposed study. The assessor is the person who will assess treatment success during follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- rESWT plus C-E drugs (Active Comparator): Patients will receive rESWT, Celecoxib and Eperisone
  Interventions: Device: rESWT; Drug: Celecoxib; Drug: Eperisone
- rESWT alone (Active Comparator): Patients will receive rESWT
  Interventions: Device: rESWT
- C-E drugs alone (Active Comparator): Patients will receive Celecoxib and Eperisone
  Interventions: Drug: Celecoxib; Drug: Eperisone

INTERVENTIONS:
Device: rESWT — rESWT will be performed as follows:
  * Four rESWT sessions
  * One rESWT session per week
  * 4 × 1000 radial extracorporeal shock waves (rESWs) per session (1000 rESWs each applied to the left and the right paravertebral muscles above L3 to S1 using the 36-mm applicator, plus 1000 rESWs each applied to the left and the right sacroiliac joint using the 15-mm convex applicator, in prone position of the patient.
  * rESWs applied at 15 Hz
  * Air pressure of the rESWT device gradually increased during the first 200 rESWs each until the maximum discomfort the patient can tolerate will be reached, followed by 800 rESWs at this air pressure / energy flux density.
  * No application of local anaesthetics
  Arms: rESWT alone; rESWT plus C-E drugs
Drug: Celecoxib — 1 x 200 mg per day for moderate pain (Numerical Rating Scale score 4-6 on an 11-point scale where 0 indicates no pain and 10 indicates worst imaginable pain), or 2 x 200 mg per day (Numerical Rating Scale 7-10), respectively, for four weeks
  Other Names: non-steroidal anti-inflammatory drug
  Arms: C-E drugs alone; rESWT plus C-E drugs
Drug: Eperisone — 3 x 50 mg per day for four weeks
  Other Names: antispasmodic drug
  Arms: C-E drugs alone; rESWT plus C-E drugs

SUMMARY:
This study tests the hypothesis that radial extracorporeal shock wave therapy (rESWT) in combination with the non-steroidal anti-inflammatory drug Celecoxib and the antispasmodic drug Eperisone (hereafter, "C-E drug therapy") is statistically significantly more effective than either rESWT or C-E drug therapy alone in the treatment of chronic non-specific low back pain.

DETAILED DESCRIPTION:
Non-specific low back pain is defined as low back pain not attributable to a recognizable, known specific pathology (e.g., infection, tumour, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome). It is second only to the common cold as the most common affliction of mankind and is among the leading complaints bringing patients to physicians' offices. The reported point prevalence of non-specific low back pain is as high as 33 percent, its one-year prevalence as high as 73 percent and its lifetime prevalence exceeds 70% in most industrialized countries, with an annual incidence of 15% to 20% in the United States of America. In physically active adults not seeking medical attention, the annual incidence of clinically significant non-specific low back pain with functional impairment is approximately 10 to 15 percent. In China, non-specific low back pain has become one of the leading causes of disability-adjusted life-years (DALYs) in 2010. Some authors reported the prevalence of non-specific low back pain as 41% in Chinese adolescents.

Management for patients with non-specific low back pain is challenged by the problems that most back pain has no recognizable cause (>85%), an underlying systemic disease is rare, and most episodes of back pain are unpreventable.

Acute non-specific low back pain (lasting three to six weeks) usually resolves in several weeks, although recurrences are common and low-grade symptoms are often present years after an initial episode. Risk factors for the development of disabling chronic or persistent non-specific low back pain (variously defined as lasting more than three months or more than six months) include preexisting psychological distress, disputed compensation issues, other types of chronic pain, and job dissatisfaction.

The goals of management for patients with non-specific low back pain are to decrease the pain, restore mobility, hasten recovery so the patient can resume normal daily activities as soon as possible, (iv) prevent development of a chronic recurrent condition, and restore and preserve physical and financial independence and comfort.

Unfortunately, few if any treatments have been proven effective for non-specific low back pain in meta-analyses, including limited bed rest, physical activity and exercise, back schools, traction, massage, chiropractic, radiofrequency denervation, paracetamol, opioids and, ultimately, surgery (in cases of cauda equina syndrome, infections, tumors and fractures compressing the spinal cord, mechanical instability of the back, and, perhaps, intractable pain with a positive straight-leg-raising test and no response to conservative therapy). Earlier studies demonstrated that muscle relaxants are effective in the management of non-specific low back pain, but the adverse effects require that they be used with caution. Accordingly, the aforementioned guideline by the American College of Physicians is only based on low- and moderate-quality evidence.

Recently extracorporeal shock wave therapy (ESWT) was introduced into the management of non-specific low back pain. The use of extracorporeal shock waves (ESWs) in medicine was first reported over 30 years ago as a treatment for kidney stones, and is commonly referred to as extracorporeal shock wave lithotripsy (ESWL). Extracorporeal shock waves are also used as a treatment for various musculoskeletal conditions such as calcifying tendinopathy of the shoulder, epicondylitis, Achilles tendinopathy and plantar fasciitis, and is commonly referred to as 'extracorporeal shock wave therapy', or 'ESWT' to differentiate from ESWL. ESWT is effective and safe, and for the aforementioned conditions randomized controlled trials (RCTs) on ESWT were the predominant type of RCT listed in the PEDro database and/or obtained the highest PEDro scores among all investigated treatment modalities.

There are three different types of ESWs used in ESWT for musculoskeletal conditions, focused, defocused and radial, and several modes of operation of focused, defocused and radial extracorporeal shock wave generators. Focused, defocused and radial ESWs are single acoustic impulses with an initial high positive peak pressure between 10 and 100 megapascals (MPa) reached in less than one microsecond (µs). The positive pressure amplitude is followed by a low tensile amplitude of a few microseconds duration that can generate cavitation. They are further characterized by a short life cycle of approximately 10-20 µs and a broad frequency spectrum. Focused ESWs differ from radial ESWs in the penetration depth into the tissue, some physical characteristics, and the technique for generating them. However, without going into detail, there is no scientific evidence in favor of either radial ESWT (rESWT) or focused ESWT (fESWT) with respect to treatment outcome, and no scientific evidence that a certain fESWT technology is superior to the other technologies.

Several molecular and cellular mechanisms were reported on how ESWs might mediate their pain-relieving action. Specifically, exposure of the distal femur of rabbits to focused ESWs decreased the amount of Substance P (SP) in the periosteum and diminished the number of neurons immunoreactive for substance P in dorsal root ganglia L5. Furthermore, application of shock waves to rat skin decreased calcitonin gene-related peptide (CGRP) immunoreactivity in dorsal root ganglion neurons. Substance P is concentrated in unmyelinated C-fibers (responsible for throbbing, chronic pain) and a subpopulation of slowly conducting, lightly myelinated A-delta nerve fibers, and is released at central and peripheral terminals of sensory nociceptive neurons after stimulation. CGRP is a marker of sensory neurons typically involved with pain perception and was immunohistochemically co-localized with substance P in capsaicin-sensitive axons. Activation of peripheral small diameter sensory neurons by local depolarization, axonal reflexes, or dorsal root reflexes releases substance P and CGRP. Both substances then act on target cells in the periphery such as mast cells, immune cells and vascular smooth muscle cells, thus producing inflammation. This phenomenon is called neurogenic inflammation, and is an inflammatory symptom that results from the release of substances from primary sensory nerve terminals. Evidence has emerged that chronic inflammation contributes to the etiology of pain in insertion tendinopathies such as tennis elbow and chronic plantar fasciitis. Furthermore, it was found that SP (as well as interleukin 1 alpha and transforming growth factor beta-1) are involved in the pathogenesis of tennis elbow, without apparent infiltration of inflammatory cells. Moreover, depletion of substance P was repeatedly shown to reduce experimentally induced inflammation of paws and joints in laboratory animals. It is therefore reasonable to hypothesize that reduction of SP and CGRP in the target tissue in conjunction with reduced synthesis of this molecule in dorsal root ganglia cells plays an important role in ESWT-mediated long-term analgesia in the treatment of musculoskeletal conditions.

With respect to non-specific low back pain it is important to note that in rats, the presence of SP and CGRP immunoreactive nerve fibers was demonstrated in the lumber facet joints. Furthermore, SP immunoreactive fibers were found more extensively in lumbar intervertebral discs from patients with discogenic low back pain than in normal control discs, together with the formation of a zone of vascularized granulation tissue from the nucleus pulposus to the outer part of the annulus fibrosus along the edges of the fissures. These findings suggested that the zone of granulation tissue with extensive innervation along the tears in the posterior part of the painful disc may be responsible for causing the pain of discography and of discogenic low back pain. Accordingly, ESWT could be of great significance in the treatment of persistent non-specific low back pain.

The studies on ESWT for non-specific low back pain performed so far have only established very limited evidence of efficacy and safety of ESWT for non-specific low back pain. This is due to low sample size, lack of power analyses, lack of reporting critical information such as the follow-up interval, and the fact that only one RCT on this indication was performed so far.

Accordingly, further research is needed to support the use of ESWT for non-specific low back pain. Taking into account the well-known molecular and cellular mechanisms of action of ESWT in pain relief (outlined in detail above), the proven efficacy and safety of rESWT for treating musculoskeletal conditions, and the fact that a ceratin rESWT device provided by Electro Medical Systems (Nyon, Switzerland) has become by far the best investigated ESWT technology in the field of Evidence Based Medicine, it is reasonable to hypothesize that treatment of non-specific low back pain with rESWT is not only effective and safe but will get widespread acceptance and clinical use as soon as effectiveness and safety will be demonstrated in a randomized controlled trial. This is the purpose of the proposed project.

The standard therapy of chronic non-specific low back pain at the Department of Pain Medicine at the First Affiliated Hospital of Zhejiang University consists of the non-steroidal anti-inflammatory drug Celecoxib and the antispasmodic drug Eperisone (hereafter, "C-E drug therapy"). Considering the established evidence of superiority of combination therapies of rESWT and other treatment modalities (such as the combination of rESWT and plantar fascia-specific stretching in case of chronic plantar fasciitis and the combination of rESWT and eccentric loading in case of chronic midportion Achilles tendinopathy) the proposed study will specifically test the hypothesis that rESWT in combination with C-E drug therapy is statistically significantly more effective than either rESWT or C-E drug therapy alone in the treatment of chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults (both male and female) with non-specific low back pain for more than three months.
* Age range: between 18 and 80 years.
* Willingness of the patient to participate in the study, and written informed consent signed and personally dated by the patient.
* Chronic non-specific low back pain clinically diagnosed as repeated lumbar sourness and swelling pain or a chronic progressive process, accompanied by (i) X-ray examination to exclude lumbar vertebrate fractures, spondylolysis, spondylolisthesis and severe osteoporosis, and/or (ii) MRI with normal signal or low nucleus pulposus signal.
* No contraindications for rESWT.

Exclusion Criteria:

* Children and teenagers below the age of 18.
* Elderly aged >80 years old
* No willingness of the patient to participate in the study, and/or written informed consent not signed and not personally dated by the patient.
* Previous spinal fracture or spinal surgery.
* Protrusion of a lumbar intervertebral disk, ankylosing spondylitis, scoliosis, lumbar spondylolisthesis and lumbar spondylolysis.
* Systemic disorders and psychiatric disorders.
* Contraindications of C-E drug treatment (treatment of patients allergy to celecoxib, eperisone or sulfonamides, patients with gastrointestinal bleeding or bleeding history, patients with renal dysfunction, patients with severe heart failure, and lactating women).
* Contraindications of rESWT ( pregnant patients, patients with blood-clotting disorders [including local thrombosis], patients treated with oral anticoagulants, patients with local tumors, patients with local bacterial and/or viral infections [including lumbar vertebral tuberculosis], and patients treated with local corticosteroid applications in the time period of six weeks before the first rESWT session [if applicable]).
* Participation in any other clinical trial in the time period of 12 weeks before potential inclusion in the proposed study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Self-Efficacy Questionnaire (PSEQ) score (Nicholas, 1989; paper presented at the annual conference of the British Psychological Society, St. Andrews, 1989) | Change from baseline PSEQ score at 12 weeks
  Patients will be asked to rate how confident they are at the time of examination despite the presence of their pain in performing the following activities:
  * I can enjoy things, despite the pain.
  * I can do most of the household chores (e.g. tidying-up, washing dishes, etc.), despite the pain.
  * I can socialize with my friends or family members as often as I used to do, despite the pain.
  * I can cope with my pain in most situations.
  * I can do some form of work, despite the pain.
  * I can still do many of the things I enjoy doing, such as hobbies or leisure activities, despite the pain.
  * I can cope with my pain without additional medication (next to rESWT plus C-E drugs, rESWT alone or C-E drugs alone, respectively).
  * I can still accomplish most of my goals in life, despite the pain.
  * I can live a normal lifestyle, despite the pain.
  * I can gradually become more active, despite the pain.

SECONDARY OUTCOMES:
Change in Numerical Rating Scale (NRS) score | Change from baseline NRS score at 2 weeks, 4 weeks, 12 weeks and 24 weeks
  The NRS will ask patients to rate their pain intensity on an 11-point scale where 0 indicates no pain and 10 indicates worst imaginable pain.
Change in Oswestry Low Back Pain Disability Questionnaire (OLDPDQ) score | Change from baseline OLDPDQ score at 2 weeks, 4 weeks, 12 weeks and 24 weeks
  The OLDPDQ score is considered the 'gold standard' of low back functional outcome tools. The questionnaire is composed of ten sections (addressing pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling); for each section the possible score is 5 and, thus, the total possible score is 50. The final score is calculated as [(sum of individual scores) / 50] *100 (%), and is interpreted as minimal disability (0% to 20%), moderate disability (21% to 40%), severe disability (41% to 60%), crippled (61% to 80%) or patients are either bed-bound or exaggerating their symptoms (81% to 100%).
Change in Patient Health Questionnaire 9 (PHQ-9) score | Change from baseline PHQ-9 score at 2 weeks, 4 weeks, 12 weeks and 24 weeks
  The PHQ-9 will be used to assess depression. Patients will be asked how often, over the last two weeks, they had been bothered by the following problems: (i) little interest or pleasure in doing things; (ii) feeling down, depressed or hopeless; (iii) trouble falling or staying asleep, or sleeping too much; (iv) feeling tired or having little energy; (v) poor appetite or overeating; (vi) feeling bad about themselves, or that they are a failure or have let themselves or their family down; (vii) trouble concentrating on things, such as reading the newspaper or watching television; (viii) moving or speaking so slowly that other people could have noticed? Or the opposite - being so fidgety or restless that they have been movin around a lot more than usual; and (ix) thoughts that they would be better of dead or of hurting themselves in some way.
Change in lumbar curvature measurements performed on lateral lumbosacral spine radiographs | Change from baseline at 12 weeks
  There is a strong relationship between non-specific low back pain and decreased lumbar lordotic curvature. Lateral X-rays of the lumbar spine will be taken in the standing position according to standard protocols in the literature, and analyzed using Cobb's angle, vertebral body and intervertebral disc wedging, and facet joint angle.
Change in Pain Self-Efficacy Questionnaire (PSEQ) score (Nicholas, 1989) | Change from baseline PSEQ score at 2 weeks, 4 weeks and 24 weeks
  Patients will be asked to rate how confident they are at the time of examination despite the presence of their pain in performing the following activities:
  * I can enjoy things, despite the pain.
  * I can do most of the household chores (e.g. tidying-up, washing dishes, etc.), despite the pain.
  * I can socialize with my friends or family members as often as I used to do, despite the pain.
  * I can cope with my pain in most situations.
  * I can do some form of work, despite the pain.
  * I can still do many of the things I enjoy doing, such as hobbies or leisure activities, despite the pain.
  * I can cope with my pain without additional medication (next to rESWT plus C-E drugs, rESWT alone or C-E drugs alone, respectively).
  * I can still accomplish most of my goals in life, despite the pain.
  * I can live a normal lifestyle, despite the pain.
  * I can gradually become more active, despite the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Zyiying Feng, MD, Principal Investigator — Department of Pain Medicine, First Affiliated Hospital of Zhejiang University, Hangzhou, China
Locations (1):
- Department of Pain Medicine, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.

REFERENCES:
- [Derived] Guo X, Li L, Yan Z, Li Y, Peng Z, Yang Y, Zhang Y, Schmitz C, Feng Z. Efficacy and safety of treating chronic nonspecific low back pain with radial extracorporeal shock wave therapy (rESWT), rESWT combined with celecoxib and eperisone (C + E) or C + E alone: a prospective, randomized trial. J Orthop Surg Res. 2021 Dec 4;16(1):705. doi: 10.1186/s13018-021-02848-x. PMID 34863239

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03337607/Prot_SAP_001.pdf